CLINICAL TRIAL: NCT05989503
Title: Initiation of Angiotensin Receptor-neprilysin Inhibitor (ARNi) and Sodium-glucose Cotransporter-2 Inhibitors (SGLT2i) in Patients With Heart Failure With Reduced Ejection Fraction (HFrEF): the INITIATE-HFrEF Randomized Open-label Trial
Brief Title: Initiation of ARNi and SGLT2i in Patients With HFrEF
Acronym: INITIATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Unidade de Investigação e Desenvolvimento Cardiovascular (UnIC) (Unknown); Rede de Investigação em Saúde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INITIATE-HFrEF; 2022-502409-14-00 (Other: EU CT Number)
Record Dates: First submitted 2023-07-14; First posted 2023-08-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Intervention Model Description: Pragmatic study to be conducted in real-life routine practice conditions with a two-arm open randomization, to evaluate the efficacy (on surrogate markers) and safety of ARNi and SGLT2i combination in patients with HFrEF/HFmrEF and the doses of ARNi.
  1. initiation of ARNi and SGLT2i simultaneously (same day or within ± 5 days);
  2. initial SGLT2i initiation followed by ARNi between week 4 and 12 after randomization.
  Assuming a primary outcome frequency of 30% in the sequential group, if there is a true difference between the intervention groups (simultaneous vs sequential) of 10%, then 62 patients are required to be 80% certain that the upper limit of a one-sided 95% confidence interval will exclude a difference in favour of the sequential group of more than 20%.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simultaneous initiation (Active Comparator): ARNi ((i.e. sacubitril/valsartan, irrespectively of brand name, at an initial dose 24/26mg b.i.d. or 49/51mg b.i.d. titrated to 97/103mg b.i.d. preferably in the first 3-6 weeks, up to 3 months of follow-up) and SGLT2i (either empagliflozin or dapagliflozin or respective combinations with other substances, providing the total dose of SGLT2i is, at least, of 10mg/d) on the same day or within ± 5 days.
  Interventions: Drug: Sacubitril-valsartan; Drug: SGLT2 inhibitor
- Sequential initiation (Active Comparator): Initial (at randomization day) SGLT2i prescription (either empagliflozin or dapagliflozin, or respective combinations with other substances, providing the total dose of SGLT2i is, at least, of 10 mg/d) followed by an ARNi initiated between weeks 4 and 12 after randomization (sacubitril/valsartan at an initial dose of 24/26mg b.i.d. or 49/51mg b.i.d., and titrated to 97/103mg b.i.d. if tolerated, according to assistant physician decision)
  Interventions: Drug: Sacubitril-valsartan; Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: Sacubitril-valsartan — Sacubitril-valsartan titration at the discretion of the treating physician
Drug: SGLT2 inhibitor — Either empagliflozin or dapagliflozin 10 mg/day

SUMMARY:
Heart failure (HF) is a condition in which the heart does not contract ("pump") or relax well, leading to insufficient perfusion of vital organs. Ankle swelling, fatigue, and breathlessness are some of the features of this syndrome. There are different causes for HF (e.g., infarct and hypertension) and two distinct types: HFpEF - HF with preserved ejection fraction - the heart "pumps" but does not relax well and HFrEF/HFmrEF - HF with reduced or mildly reduced ejection fraction - where the heart does not "pump" properly, here referred to as having HFrEF.

Patients with HFrEF experience substantially shorter life expectancies compared with people in the general population of similar age. Compared to the different available therapeutics for HFrEF patients, angiotensin receptor-neprilysin inhibitor (ARNi), sacubitril/valsartan, has shown superiority for improving clinical outcomes. Furthermore, the new recently drug sodium-glucose cotransporter 2 inhibitor (SGLT2i) was proven to reduce mortality and morbidity on top of well-adapted background therapy.

This work aims to test the safety of ARNi and SGLT2i initiation by comparing a strategy of simultaneous initiation of ARNi and SGLT2i versus sequential initiation of a SGLT2i first followed by an ARNi.

DETAILED DESCRIPTION:
Sacubitril/valsartan and SGLT2i reduced HF hospitalizations and mortality in patients with heart failure and a reduced ejection fraction with a rapid onset of action, but the timing of initiation of each drug is uncertain. Clinicians may be reluctant to initiate both therapies simultaneously due to fear of adverse events (e.g., hypotension and worsening renal function) which may delay the initiation of (at least one) of these life-saving therapies.

This study aims to fill this gap in knowledge by studying the initiation of sacubitril/valsartan and a SGLT2i simultaneously or in sequence. This study will better inform clinicians on their daily decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Heart failure symptoms (NYHA II, III or IV)
3. Left ventricle ejection fraction ≤ 49% (assessed by transthoracic echocardiogram)
4. Glomerular filtration rate ≥ 25 ml/min/1.73m2 (CKD-EPI formula)
5. Serum potassium (K+) ≤ 5.4 mmol/L
6. Systolic blood pressure ≥ 100 mmHg
7. Not treated with ARNi nor with SGLT2i within the previous month (30 days before inclusion, except if initiated 5 days before randomization; patients treated with an ACEi or ARB can be included and maintain their therapy until the switch to an ARNi is performed)
8. If female, she must not be a woman of childbearing potential. That is, she must be:

   1. Surgically sterilized (e.g., underwent hysterectomy, bilateral salpingectomy or bilateral oophorectomy)
   2. Clinically diagnosed infertile
   3. In a post-menopausal state, defined as no menses for 12 months without an alternative medical cause
9. If female patient of childbearing potential, she must have a negative serum pregnancy test at Visit 1 (Day 0) and must agree to consistently and correctly use (from 28 days prior to first study treatment administration until at least 7 days after last study treatment administration) one of the following highly effective methods of contraception:

   1. Abstinence of heterosexual intercourse (when this is in line with preferred and usual lifestyle of the subject)
   2. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
   3. Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
   4. Intrauterine device
   5. Intrauterine hormone-releasing system
   6. Bilateral tubal occlusion
   7. Vasectomized partner, who has received medical assessment of the surgical success, or clinically diagnosed infertile partner

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site)
2. Participation in another clinical study with an investigational product during the last month
3. Unwilling to sign inform consent
4. Patients with a known hypersensitivity or intolerance to ARNi or SGLT2i or any of the excipients of the products
5. Hospitalization due to non-cardiovascular causes, surgical procedure, coronary, cerebral or peripheral vascular events or sepsis in the prior month
6. Cancer (life limiting with an estimated life expectancy of less than 2 years based on investigator's judgement)
7. Previously confirmed cardiac amyloidosis
8. History of angioedema
9. Implantable cardioverter-defibrillators or cardiac resynchronization therapy within 3 months prior to screening or if there is an intent to implant either device in the 3 months following screening
10. Female patients currently pregnant (confirmed by a positive pregnancy test) or intent to become pregnant or breast feeding
11. Severe valvulopathy according to the echocardiogram report
12. Previous history of ketoacidosis due to SGLT2i

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Composite outcome (time-to-first event' occurrence during the 6 months of follow-up): | visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  * Symptomatic hypotension (systolic blood pressure <100 mmHg with signs or symptoms compatible with hypoperfusion);
  * Hyperkalaemia (serum potassium >6.0 mmol/L);
  * Hypokalemia (serum potassium <3.0 mmol/L);
  * eGFR drop ≥50% from baseline or eGFR <15 ml/min/1.73m2 or renal transplant or dialysis;
  * Increase in diuretic dose due to worsening heart failure;
  * Use of intravenous diuretics for worsening heart failure;
  * Heart failure hospitalization;
  * Death from cardiovascular causes.

SECONDARY OUTCOMES:
Symptomatic hypotension (systolic blood pressure <100 mmHg with signs or symptoms compatible with hypoperfusion) | visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Time to event' occurrence during the 6 months of follow-up
Hyperkalaemia (serum potassium >6.0 mmol/L) | visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Time to event' occurrence during the 6 months of follow-up
Hypokalemia (serum potassium <3.0 mmol/L) | visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Time to event' occurrence during the 6 months of follow-up
eGFR drop ≥50% from baseline or eGFR <15 ml/min/1.73m2 or renal transplant or dialysis | visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Time to event' occurrence during the 6 months of follow-up
Increase in diuretic dose due to worsening heart failure | visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Time to event' occurrence during the 6 months of follow-up
Use of intravenous diuretics for worsening heart failure | visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Time to event' occurrence during the 6 months of follow-up
Heart failure hospitalization | visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Time to event' occurrence during the 6 months of follow-up
Death from cardiovascular causes | visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Time to event' occurrence during the 6 months of follow-up
NT-pro BNP or BNP (log) | visit 1 (day 0); visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
High sensitivity C-reactive protein | visit 1 (day 0); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
Atrial fibrillation/flutter | visit 1 (day 0); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Electrocardiogram (yes/no)
Systolic and diastolic blood pressure | visit 1 (day 0); visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Measure in the clinical appointments
High sensitivity Troponin | visit 1 (day 0); visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
Left atrial volume | visit 1 (day 0); visit 4 (visit 3 + 90±15 days)
  Transthoracic echocardiogram
Left ventricular systolic volume | visit 1 (day 0); visit 4 (visit 3 + 90±15 days)
  Transthoracic echocardiogram
Left ventricular diastolic volume | visit 1 (day 0); visit 4 (visit 3 + 90±15 days)
  Transthoracic echocardiogram
LV mass | visit 1 (day 0); visit 4 (visit 3 + 90±15 days)
  Transthoracic echocardiogram
LV ejection fraction | visit 1 (day 0); visit 4 (visit 3 + 90±15 days)
  Transthoracic echocardiogram
Pulmonary artery systolic pressure | visit 1 (day 0); visit 4 (visit 3 + 90±15 days)
  Transthoracic echocardiogram
Serum sodium | visit 1 (day 0); visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
Serum potassium | visit 1 (day 0); visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
Serum creatinine | visit 1 (day 0); visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
Glomerular filtration rate (eGFR) | visit 1 (day 0); visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Calculated from the serum creatinine using the 2021 CKD-EPI creatinine-based formula
Urinary sodium | visit 1 (day 0); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Spot urine sample
Urinary potassium | visit 1 (day 0); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Spot urine sample
Microalbuminuria | visit 1 (day 0); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Spot urine sample
Total Cholesterol | visit 1 (day 0); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
LDL Cholesterol | visit 1 (day 0); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
HDL Cholesterol | visit 1 (day 0); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
Triglycerides | visit 1 (day 0); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
Glucose | visit 1 (day 0); visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Measured in blood samples
Glycated hemoglobin (HbA1C) | visit 1 (day 0); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
Uric acid | visit 1 (day 0); visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
TSH | visit 1 (day 0); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
Free thyroxin | visit 1 (day 0); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
ALAT | visit 1 (day 0); visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
ASAT | visit 1 (day 0); visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
Gamma-GT | visit 1 (day 0); visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
Alkaline Phosphatase | visit 1 (day 0); visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
Total bilirubin | visit 1 (day 0); visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
Serum iron | visit 1 (day 0); visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
Ferritin | visit 1 (day 0); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
Transferrin saturation | visit 1 (day 0); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Concentration measured in blood samples
Functional class (NYHA, New York Heart Association) | visit 1 (day 0); visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  Assessed by the medical doctors in the clinical appointments (I / II / III / IV)
Quality of life (KCCQ, Kansas City Cardiomyopathy Questionnaire) | visit 1 (day 0); visit 3 (visit 2 + 60 ±15 days); visit 4 (visit 3 + 90±15 days)
  HR-QoL assessed by the Kansas City Cardiomyopathy Questionnaire a 12-item instrument. All items are measured on a Likert scale with 5-7 response options. KCCQ scores are scaled from 0 to 100 and summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent
Dosage titration of sacubitril/valsartan up to the dose 97/103 mg (b.i.d.) at 3 months | visit 2 (day 23 to 37); visit 3 (visit 2 + 60 ±15 days)
  Assessed by the medical doctors in the clinical appointments

CONTACTS AND LOCATIONS:
Overall Officials: João P. Ferreira, MD, PhD, Principal Investigator — Universidade do Porto
Locations (5):
- Portugal (5):
  - Centro Hospitalar Universitário de Santo António, Porto, Porto District
  - Centro Hospitalar Universitário São João, Porto
  - Faculty of Medicine (FMUP), Porto
  - Centro Hospitalar Vila Nova de Gaia/Espinho, Porto
  - Unidade Local de Saúde de Matosinhos - Hospital Pedro Hispano, Porto